CLINICAL TRIAL: NCT05710406
Title: Randomized Trial of Consolidation Targeted Adjuvant Therapy With Encorafenib and Cetuximab Versus Usual Care for Patients With Stage II/III BRAF V600E Colon Cancer
Brief Title: Testing the Use of BRAF-Targeted Therapy After Surgery and Usual Chemotherapy for BRAF-Mutated Colon Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A022004; NCI-2022-09129 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Colon Adenocarcinoma; Microsatellite Stable Colon Carcinoma; Stage IIB Colon Cancer AJCC v8; Stage IIC Colon Cancer AJCC v8; Stage III Colon Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms | interventions — encorafenib; Cetuximab; Magnetic Resonance Spectroscopy; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (encorafenib, cetuximab) (Experimental): Patients receive encorafenib PO and cetuximab IV on study. Patients also undergo collection of blood samples throughout the study and CT or MRI during screening and follow-up.
  Interventions: Drug: Encorafenib; Biological: Cetuximab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm II (patient observation) (Active Comparator): Patients undergo observation per usual care on study. Patients also undergo collection of blood samples throughout the study and CT or MRI during screening and follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Patient Observation

INTERVENTIONS:
Drug: Encorafenib — Given PO
  Other Names: Braftovi; LGX-818
  Arms: Arm I (encorafenib, cetuximab)
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar KL 140; Chimeric Monoclonal Antibody C225; Erbitux
  Arms: Arm I (encorafenib, cetuximab)
Procedure: Biospecimen Collection — Undergo collection of blood samples
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Other: Patient Observation — Undergo observation per usual care
  Other Names: Watchful Waiting
  Arms: Arm II (patient observation)

SUMMARY:
This phase II/III trial compares treatment with encorafenib and cetuximab to usual care (patient observation) for reducing the chance of cancer recurrence after standard surgery and chemotherapy in patients with BRAF-mutated stage IIB-III colon cancer. Encorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cetuximab is in a class of medications called monoclonal antibodies. It binds to a protein called EGFR, which is found on some types of tumor cells. This may help keep tumor cells from growing. Giving encorafenib and cetuximab after standard surgery and chemotherapy may be more effective at reducing the chance of cancer recurrence compared to the usual patient observation.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

I. To evaluate and compare 6 month circulating tumor deoxyribonucleic acid (ctDNA) clearance rate in study patients with detectable ctDNA prior to randomization to targeted BRAF therapy versus usual care after standard adjuvant chemotherapy. (Phase II) II. To evaluate and compare 6 month ctDNA recurrence-free survival (ctDNA-RFS) rate in study patients with undetectable ctDNA prior to randomization to targeted BRAF therapy versus usual care after standard adjuvant chemotherapy. (Phase II) III. To evaluate and compare disease-free survival (DFS) (measured from randomization) in patients with resected stage III or high-risk (pT4) stage II mismatch repair protein (MMR) proficient BRAF V600E colon cancer treated with targeted BRAF therapy versus usual care after standard adjuvant chemotherapy. (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate and compare overall survival (OS) between the two treatment arms.

II. To evaluate and compare the toxicity profile between the two treatment arms.

III. To evaluate and compare the alternative DFS endpoint (measured from date of primary tumor resection) between the two treatment arms.

IV. To evaluate and compare DFS in the subset of patients with detectable ctDNA prior to randomization between the two treatment arms.

EXPLORATORY OBJECTIVE:

I. To evaluate and compare patient-reported outcomes for symptoms of rash, diarrhea, and fatigue according to Patient Reported Outcomes Version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) between the two treatment arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive encorafenib orally (PO) and cetuximab intravenously (IV) on study. Patients also undergo collection of blood samples throughout the study and computed tomography (CT) or magnetic resonance imaging (MRI) during screening and follow-up.

ARM II: Patients undergo observation per usual care on study. Patients also undergo collection of blood samples throughout the study and CT or MRI during screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION (STEP 0) ELIGIBILITY CRITERIA:
* BRAF V600 mutational status may be determined either locally or by central testing. This testing is mandatory prior to registration to determine eligibility. Tissue submission should be initiated as soon after surgery as possible. For tumors evaluated at local laboratories, formalin-fixed paraffin-embedded (FFPE) tumor tissue must still be submitted for central confirmation of BRAF status
* REGISTRATION (STEP 1) ELIGIBILITY CRITERIA:
* Histologically-proven stage III (any T [Tx, T1, T2, T3, or T4], N1-2M0; includes N1C) or high-risk (pT4) stage II colon adenocarcinoma. Tumors must be deemed to originate in the colon including tumors that extend into/involve the small bowel (e.g. those at the ileocecal valve) and must have been completely resected
* BRAF V600E mutation
* MMR proficient (pMMR) or microsatellite stable (MSS) tumor
* Histologic documentation: adenocarcinoma
* Stage: III (any T [Tx, T1, T2, T3, or T4], N1-2M0; includes N1C) or high-risk II (pT4)
* Tumor site: colon
* Patients must have received at least 3 months of adjuvant chemotherapy with either leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX) (minimum of 5 cycles) or capecitabine and oxaliplatin (CAPOX) (minimum of 3 cycles)
* Adjuvant therapy must be completed at most 8 weeks prior to registration
* No other prior medical therapy (chemotherapy, immunotherapy, biologic, or targeted therapy) or radiation therapy for the current colon cancer is permitted
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelet count >= 75 x 10^9/L
* Hemoglobin > 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x ULN
* Corrected QT (QTc) Interval =< 480 msec
* Creatinine = calculated (calc.) creatinine clearance >= 40 mL/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* No medical condition such as uncontrolled infection, uncontrolled diabetes mellitus, or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Patients with known history or current symptoms of cardiac disease or history of treatment with cardiotoxic agents in the last 12 months, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* No uncontrolled or poorly-controlled hypertension (> 180 mmHg systolic or > 130 mmHg diastolic)
* No history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab
* No "currently active" second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 3 years

  * Patients are not considered to have a "currently active" malignancy if they had a gastric or bowel carcinoid < 1 cm, ductal carcinoma in situ (DCIS)/lobular carcinoma in situ (LCIS) of the breast without invasive cancer, or endometrial dysplasia/carcinoma in situ
  * Patients are not considered to have a "currently active" malignancy if they had a sebaceous neoplasm (sebaceous adenoma, sebaceous epithelioma, sebaceous adenocarcinoma, keratoacanthoma, and squamous cell carcinoma) that was noninvasive
* No known medical condition causing an inability to swallow oral formulations of agents
* No residual Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 grade >= 2 toxicity from prior chemotherapy, with the exception of grade 2 alopecia or neuropathy
* Drugs that prolong the QTc interval should be avoided if possible, as encorafenib can prolong the QTc interval. Drugs that are generally accepted to have a risk of causing Torsades de Pointes should be discontinued or replaced with drugs that do not carry this risk if at all possible. Patients who receive potential QTc-prolonging medications should be monitored closely
* Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed during treatment on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study
* Chronic concomitant treatment with strong CYP3A4 inducers is not allowed during treatment on this study. Patients must discontinue the drug 14 days prior to registration on the study

Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2034-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor deoxyribonucleic acid (ctDNA) clearance rate (Phase II; ctDNA positive cohort) | At 6 months after randomization
  defined as the proportion of patients with undetectable ctDNA status at 6 months after randomization among patients with detectable ctDNA status at randomization. The ctDNA clearance rate at 6 months after randomization in experimental arm will be compared to control arm by Chi-squared test. The one-sided p-value will be reported. Due to small sample size, Cochran and Mantel-Haenszel test, stratified by stratification factors will be performed as sensitivity analysis.
tDNA recurrence-free survival rate (ctDNA-RFS) (Phase II; ctDNA negative cohort) | at 6 months after randomization
  Defined as the proportion of patients who remained undetectable ctDNA status, recurrence-free, and alive at 6 months after randomization among patients with undetectable ctDNA status at randomization. The ctDNA-RFS in experimental arm will be compared to control arm by Cochran and Mantel-Haenszel test, stratified by stratification factors. The one-sided p-value will be reported.
Disease free survival (DFS) (Phase III) | Assessed up to 6 years after randomization
  Defined as the time from the date of randomization to the date of first documented recurrence or death due to all cause, whichever occurs first. Patients without events observed at the end of the study will be censored at the date of last disease evaluation which shows no evidence of disease. At each analysis (Interim #1, Interim #2, and Final), stratified Cox model will be conducted to compare DFS in the experimental arm to DFS in the control arm with stratification factors as stratum, based on all data collected at the analysis time point.

SECONDARY OUTCOMES:
Overall Survival | Assessed up to 6 years
  Defined as the time from the date of randomization to death due to all causes. The distributions of time-to-event endpoints will be estimated, in each arm, using the method of Kaplan-Meier and compared by a stratified Cox regression model.
Incidence of adverse events after randomization | up to 6 years
  The maximum grade for each type of adverse events that are possibly, probably, or definitely related to study treatments will be summarized for each patient. The frequency tables will be reviewed to determine the patterns. The overall adverse event rates for grade 4 or higher adverse events will be compared between two treatment groups using Chi-square test (or Fisher's exact test if the data in the contingency table is sparse).
Alternative disease free survival | assessed up to 6 years
  Defined as the time from the date of primary tumor resection to the date of first documented recurrence or death due to all cause, whichever occurs first. The distributions of time-to-event endpoints will be estimated, in each arm, using the method of Kaplan-Meier and compared by a stratified Cox regression model.

OTHER OUTCOMES:
• Patient Reported Outcomes Version of Common Terminology Criteria for Adverse Events for symptoms of rash, diarrhea, and fatigue | up to 6 years
  summarized for each patient.

CONTACTS AND LOCATIONS:
Locations (202):
- United States (202):
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided